CLINICAL TRIAL: NCT03951844
Title: Wearability, Saefty and Usability Assessment for the Upper Limb Exoskeleton BRIDGE/EMPATIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alessandra Pedrocchi (Other)
Responsible Party: Sponsor-Investigator, Alessandra Pedrocchi, Professor, Politecnico di Milano
Organization: Politecnico di Milano (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GIP-530
Record Dates: First submitted 2019-05-13; First posted 2019-05-15 (Actual); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Muscular Dystrophies
Keywords: Exoskeleton; Upper limb; Assistive device
MeSH Terms: conditions — Muscular Dystrophies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Each participant is evaluated while wearing or not wearing the device.
  Interventions: Device: BRIDGE/EMPATIA exoskeleton

INTERVENTIONS:
Device: BRIDGE/EMPATIA exoskeleton — The participant wears the exoskeleton on his/her left arm, and he/she controls it by means of a joystick or vocal commands.

SUMMARY:
The study is a feasibility study or pilot study, that is a clinical investigation to acquire the preliminary information on a motorized exoskeleton (BRIDGE / EMPATIA exoskeleton) for the movement of the upper limb in order to develop it, including design changes. The primary objective of the clinical trial is to assess the fit, safety and usability of the device in supporting the execution of daily activities for patients suffering from muscular dystrophy. The risk analysis for the BRIDGE / EMPATIA device does not present particular criticalities that preclude the use of the device in the target population. In any case, during the trial eventual adverse events are recorded for the verification of safety..

ELIGIBILITY:
Inclusion criteria:

1. Availability of the patient and/or caregiver at the signing of the informed consent for participation in a clinical trial study protocol
2. Defined diagnosis of Muscular Dystrophy (Duchenne, Becker, Cingoli type 2 and facio-scapulo-humeral). Biopsy will not be performed except in cases where a diagnostic need arises.
3. Wheelchair bounded
4. Significant weakness in the muscular districts of the shoulder girdle and the proximal upper limb portion detected by the MRC scale (between 0 and 2)
5. Cognitive skills that allow the understanding and management of the device
6. Arm length measured from the shoulder to the elbow between 26.5 cm and 28.7 cm; forearm length, measured between elbow and wrist, maximum 22.4 cm

Exclusion criteria:

1. Presence of important comorbidities (epilepsy, dependence 24/24 hours from non-invasive and invasive ventilation)
2. Behavioral and psychiatric disorders (e.g., emotional problems, depression)
3. Inability to maintain a sitting position in a wheelchair

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-06-26 (Actual); Primary Completion 2019-04-02 (Actual); Study Completion 2019-04-02 (Actual)

PRIMARY OUTCOMES:
Performance of Upper Limbs scale (PUL) | Change from baseline PUL without the exoskeleton and PUL wearing the exoskeleton within 15 days.
  The PUL includes 22 items with an entry item to define the starting functional level and 21 items subdivided into shoulder level (4 items), middle level (9 items) and distal level (8 items). For weaker patients, a low score on the entry item means high-level items do not need to be performed. Each dimension can be scored separately with a maximum score of 16 for the shoulder level, 34 for the middle level and 24 for the distal level. A total score can be achieved by adding the three level scores, with a maximum global score of 74. The lower the score, the higher the disability.
  Pane et al., Reliability of the Performance of Upper Limb assessment in Duchenne muscular dystrophy, Neuromuscular disorders 2014, 24:201-206.

SECONDARY OUTCOMES:
ABILHAND | Change from baseline PUL without the exoskeleton and PUL wearing the exoskeleton within 15 days.
  Self-administered questionnaire aimed at measuring manual ability in daily life. Patients are asked to answer 14 questions plus 4 items differentiated with respect to the age of participant (older or younger than 15 years). Overall, the Abilhand questionnaire has 22 items. For each item, the participant has to answer if the presented action is "impossible", "difficult" or "easy" to be performed in his/her opinion. A three-level scale is used to calculate a total score according to the answer given: "impossible" (0 points), "difficult" (1 point) and "easy" (2 points). The higher the score, the easier the perception of self-ability. Data are converted to a probabilistic model through the Rasch model, which estimates the item difficulty and a patient's manual ability on a standard linear scale, within a probabilistic framework.
  Penta et al., ABILHAND: a Rasch-built measure of manual ability, Archives of Physical Medicine and Rehabilitation 1998, 79:1038-1042.
Technology acceptance model (TAM) questionnaire | Within 15 days from the baseline
  The technology acceptance model (TAM) is an information systems theory that models how users come to accept and use a technology. A dedicated TAM has been developed, and administered to the patients in the form of 26 questions on the evaluation of different aspects of the device (e.g., saefty, confort, etc.). For each item, the patient has to provide a score from 1 to 5, where 1 is completely disagree and 5 is completely agree. The higher the score, the better the technology acceptance.
System usability scale (SUS) | Within 15 days from the baseline
  It is a ten-items scale giving a global view of subjective assessments of usefulness as a combination of effectiveness, efficiency, and satisfaction. Each item score contribution ranged from 1 to 5. For items 1, 3, 5, 7 and 9 (the positively worded items) the score contribution was the scale position given by the subject minus 1. For items 2, 4, 6, 8 and 10 (the negatively worded items), the contribution was equal to 5 minus the scale position. Then, the scores were summed and multiplied by 2.5 to obtain the overall value of SUS. Scores can range from 0 to 100. SUS is evaluated according to Bangor research guidelines (Bangor et al., An Empirical Evaluation of the System Usability Scale, International Journal of Human-Computer Interaction, 2008, 24:574-594): scores in the ranges [55, 75], [75.1, 87.5] and [87.6, 100] indicated respectively "good", "excellent" and "very excellent".
  Brooke, SUS - A quick and dirty usability scale, Usability evaluation in industry, 1996, 194:4-7.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - IRCCS E. Medea - La Nostra Famiglia, Bosisio Parini, LC
  - Villa Beretta, Costa Masnaga, LC

IPD SHARING:
Plan to Share IPD: Undecided